CLINICAL TRIAL: NCT00997867
Title: Perineural Catheter Insertion Distance for Continuous Peripheral Nerve Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Brian Ilfeld, M.D., M.S./Principal Investigator, University of California, San Diego, Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Catheter Insertion Distance
Record Dates: First submitted 2009-10-18; First posted 2009-10-19 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Lower Extremity Surgery; Upper Extremity Surgery; Post-operative Pain
Keywords: Pain; Surgery; Catheter; Nerve Block; Popliteal; Sciatic; Femoral; Interscalene; UCSD; Moderate-to-severe pain; Perineural Catheter; Orthopedic Surgery
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Catheter 0-1cm past needle tip (Active Comparator): Patients will be receiving a sciatic (popliteal), femoral, or interscalene nerve block and will be randomized to having the catheter placed 0-1cm past the needle tip. The patient will be called the following day by research staff to assess their post-surgical pain.
  Interventions: Procedure: Sciatic catheter left 0-1cm past needle tip vs. 5-6cm past needle tip
- Catheter placed 5-6cm past needle tip (Active Comparator): Patients will be receiving a sciatic (popliteal), femoral, or interscalene nerve block and will be randomized to having the catheter placed 5-6cm past the needle tip. Patients will be called the following day by research staff to assess their post-surgical pain.
  Interventions: Procedure: Sciatic catheter left 0-1cm past needle tip vs. 5-6cm past needle tip

INTERVENTIONS:
Procedure: Sciatic catheter left 0-1cm past needle tip vs. 5-6cm past needle tip — Patients undergoing orthopedic surgery who are getting a perineural catheter will be randomized to one of two groups: catheter tip placed 0-1cm past needle tip or catheter tip placed 5-6cm past needle tip. Patients will be called by research staff the day following surgery to assess their post-surgical pain using a numeric rating scale.

SUMMARY:
This is a research study to determine if the effects of continuous peripheral nerve blocks are influenced by the distance of insertion past the needle tip of the perineural catheter.

DETAILED DESCRIPTION:
Specific Aim: Research study to determine the relationships between perineural catheter insertion distance and subsequent continuous peripheral nerve block effects.

Hypothesis: during ultrasound-guided perineural catheter placement, inserting the catheter 0-1cm past the needle tip is associated with decreased postoperative pain compared with inserting the catheter 5-6cm past the needle tip.

ELIGIBILITY:
Inclusion Criteria:

* undergoing surgery with a planned popliteal perineural catheter for postoperative analgesia
* age 18 years or older

Exclusion Criteria:

* pregnancy
* inability to communicate with the investigators and hospital staff
* incarceration
* clinical neuropathy in the surgical extremity
* chronic high-dose opioid use
* history of opioid abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Average pain in the three hours previous to a phone call the day following surgery as measured on a numeric rating scale (0-10, 0=no pain, 10=worst imaginable pain). | Day 1 after surgery, 3 hours prior to phone call

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States